CLINICAL TRIAL: NCT04985669
Title: Study of Comparative Effectiveness of Prucalopride and Lubiprostone in Constipation Predominant Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Sandip Kumar Bhowmick, Principle investigator, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3420
Record Dates: First submitted 2021-07-12; First posted 2021-08-02 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — prucalopride

STUDY DESIGN:
Intervention Model Description: Quasi experimental
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- prucalopride group (Experimental): prucalopride group will receive prucalopride 2 mg once daily
  Interventions: Drug: Prucalopride 2mg
- Lubiprostone group (Active Comparator): lubiprostone group will receive lubiprostone 8 microgram twice daily
  Interventions: Drug: Prucalopride 2mg

INTERVENTIONS:
Drug: Prucalopride 2mg — one group of patient will receive prucalopride once daily one group of patient will receive lubiprostone twice daily
  Other Names: calopride

SUMMARY:
This will be a semi-experimental study on constipation predominant IBS patient. One group of patient will receive prucalopride 2mg daily and another group of patient will receive lubiprostone 8 microgram twice daily. IBS-SSS and IBS-QOL score will be recorded at baseline and at follow up at 3 week and 6 week. Effectiveness of both drug will be evaluated by comparing the baseline data with data at 3 week and 6 week(IBS-SSS and IBS-QOL).

DETAILED DESCRIPTION:
Consecutive patients of both sexes age between 18-50 years attended the outpatient department of Gastroenterology, BSMMU, meeting the inclusion Criteria entered a 2 week screening period. During this period, patients were required to discontinue all laxative medications. All participants will be advised to maintain a stable diet with no significant changes in their consumption of liquids or fiber or in their level of physical activity.

During the screening period, patients accessed and diary system on a daily basis to report the occurrence and time of all spontaneous bowel movements (SBMs), defined as those that occurred without the use of rescue medications. If the patient did not experience a SBM for 3 or more consecutive days and needed relief, the study investigator could authorize the patient to administer a rescue medication. Initial rescue treatment consisted of a 10 mg bisacodyl. If this was not successful a Fleet enema could then be used. If both of these treatment options were unsuccessful, an alternative medication could be prescribed after consultation with the investigator. At the end of the screening period, patients were assessed by medical history, physical examination, and laboratory tests (CBC, ESR, CRP, RBS, S. creatinine, S.TSH and ECG) will be done. ECG will be done from cardiology OPD, BSMMU, and rest of the investigations from Department of Laboratory Medicine, BSMMU. Report will be noted in the standard data sheet. Any alternative diagnosis if proven by clinical examination or laboratory investigation will be excluded from the study

The subject will be recruited according to sample size. Selection into two groups will be performed non probability sampling method. An independent treatment codes and allocation will be maintained. Patients enrolled in trial were selected to receive either or prucalopride 2 mg once daily at morning before breakfast or lubiprostone 8 mcg twice daily after meal. Before starting treatment each individual will undergo a baseline assessment during which demographic data, IBS symptoms and QOL data will be recorded. Each drug was administered after with at least 8 ounces of water for a period of 6 weeks. A reduction to once-daily dosing was allowed, at the discretion of the investigator, if the patient experienced nausea or diarrhea for more than 2 days or if patients experienced other adverse events. During treatment, patients were prohibited from taking prescription or OTC medications for constipation.

Non constipation-related prescriptions and other OTC medications were allowed and their usage was documented as was as any medication change. As in the screening period, the use of rescue medications was allowed in those who failed to have a spontaneous bowel movement for 3 or more consecutive days and thus needed relief. During the 6-week study phase, clinic visits were conducted at weeks 3 and 6 week and phone interviews were performed at 1 week after starting and 2 week after the end at study period. At each clinic visit, the daily diary information was reviewed and discussed with the patient, adverse events were recorded, remaining capsules were collected to assess compliance and assessments of vital signs and laboratory parameters were performed. Patients also completed the IBS-QOL and IBS-SSS at week 3 and 6 visits. Patients will be asked to return with the strips of the ingested drugs at the end of the treatment to count & ensure compliance. Any adverse effect due to drugs will also be noted at the same time.

IBS-SSS is a 5 item tools. It is primarily a measure of IBS symptoms including abdominal pain and distension as well as bowel satisfaction. This scale evaluates IBS symptoms: abdominal pain, abdominal distension, stool frequency and consistency and interference with life in general. The IBS-SSS calculates the sum of these 5 items scored on a visual analogue scale from 0-100. Determination of severity of each symptoms is determined by patient. The nature of the items on IBS-SSS is appropriate to be used in clinical trials. The items are summed and thus the total score can range from 0 to 500 points. IBS severity has the following defined ranges: mild 75-174, moderate 175-300, and severe > 300

The IBS-QOL questionnaire is a 34-item instruments which assess QOL impairment due to IBS symptoms. Each item is scored on a five-point scale (1 = not at all, 5 = a great deal) that represents one of eight dimensions (dysphoria, interference with activity, body image, health-related worries, food avoidance, social reactions, sexual dysfunction, and relationships). Items are scored to derive an overall total score of IBS related QOL. To facilitate score interpretation, the summed total score is transformed to a 0-100 scale ranging from zero (poor QOL) to 100 (maximum QOL). The QOL instrument will be given to each patient before treatment is started; the patient will complete the form according to schedule and all data will be recorded and entered onto a data sheet.

ELIGIBILITY:
Inclusion criteria:

* Meet Rome IV criteria for IBS-C
* Patients given informed written consent

Exclusion Criteria:

* Current treatment with laxative or SSRI
* Use of any medication indicated for treatment of IBS within preceding 2 weeks of enrollment
* Organic disorder of the large or small bowel (e.g. inflammatory bowel disease, tuberculosis, diverticular disease)
* Diagnosis of any medical condition associated with constipation except IBS-C (e.g DM, Hypothyroidism, CVD, parkinsonism)
* Clinical feature suggestive of organic disease (e.g. unexplained significant weight loss, rectal bleeding)
* Previous gastrointestinal or abdominal surgery (except for common causes unrelated to IBS)
* Abnormal laboratory tests (CBC, CRP, RBS, S. Creatinine, S.TSH, ECG)
* Mechanical obstruction
* Known severe depression, psychiatric disorder.
* Pregnancy or lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change in Irritable Bowel Syndrome-Symptom Severity Score (IBS-SSS score), range from 0 to 500, higher scores mean worse outcome | 6 weeks
  Change in Irritable Bowel Syndrome-Symptom Severity Score (IBS-SSS score) compared to baseline

SECONDARY OUTCOMES:
Change in Irritable Bowel Syndrome-Quality of Life (IBS -QOL score), range from 0 to 100, higher scores mean worse outcome | 6 weeks
  Change in Irritable Bowel Syndrome-Quality of Life (IBS -QOL score) compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Suitana Meftaul Jannat, MBBS, Principal Investigator — Resident Doctor
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No